CLINICAL TRIAL: NCT03421925
Title: Effects of Using Divided Mesh and Using a Non Divided Mesh on Testicular Blood Flow and Volume in Laparoscopic Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Murat Ferhat Ferhatoglu, Assistant Professor, M.D., Okan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OkanU
Record Dates: First submitted 2018-01-26; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Divided mesh group (Other): In this group, surgeon will use a mesh divided in to two legs in laparoscopic totally extraperitoneal repair
  Interventions: Procedure: Laparoscopic totally extraperitoneal procedure for inguinal hernia
- Non divided mesh group (Other): In this group, surgeon will use a non divided mesh in laparoscopic totally extraperitoneal repair
  Interventions: Procedure: Laparoscopic totally extraperitoneal procedure for inguinal hernia

INTERVENTIONS:
Procedure: Laparoscopic totally extraperitoneal procedure for inguinal hernia — Laparoscopic totally extraperitoneal procedure for inguinal hernia is a technique that is done by not entering the peritoneal cavity

SUMMARY:
Laparoscopic inguinal hernia repair techniques has been compared with the open techniques in several studies. However, no one studied about the different uses of the same type of mesh on the same surgical technique, and effects of this different use on testicular volume and blood flow. The objective of this study is to investigate the effects at 6 months of the divided and non divided mesh in laparoscopic totally extraperitoneal hernia repair technique on testicular volume and blood flow by use of Doppler Ultrasonography

ELIGIBILITY:
Inclusion Criteria:

Patients with unilateral inguinal hernia Male patients

-

Exclusion Criteria:

Patients have femoral hernia Patients have bilateral inguinal hernia Patients have recurrent inguinal hernia Female patients Patients with history of pelvic surgery Patients with history of pelvic major trauma Patients with history of pelvic radiotherapy Patients have previous scrotal trauma or surgery history Patients have heavy cardiac diseases, pulmonary diseases Patients have benign prostate hyperplasia Patients have history of incarceration of inguinal hernia

-

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — In this study, we are going to measure parameters about testicles.
Enrollment: 150 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2019-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Testicular volume | 6 months

SECONDARY OUTCOMES:
Testicular artery blood flow | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Okan University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No